CLINICAL TRIAL: NCT04427163
Title: Assesment of Multiomics Profiles in Health and Disease - Corelation with the Disease Phenotype.
Brief Title: Assesment of Multiomics Profiles in Health and Disease.
Acronym: ENIGMA
Status: Recruiting | Type: Observational
Sponsor: The Institute of Molecular and Translational Medicine, Czech Republic (Other)
Responsible Party: Sponsor
Other Study IDs: 302
Record Dates: First submitted 2020-04-16; First posted 2020-06-11 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Genetic Predisposition to Disease
Keywords: genomic profile; disease phenotype; proteomic profile; metabolomic profile; transcriptomic profile
MeSH Terms: conditions — Genetic Predisposition to Disease | interventions — Health Status; alpha-methylacyl-CoA racemase; Ethnicity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Genomic, transcriptomic, proteomic, metabolomic profiles: Determination of genomic, transcriptomic, proteomic, metabolomic profiles in subjects.
  Interventions: Genetic: Blood sample analysis; Other: Health status; Other: Race and ethnicity

INTERVENTIONS:
Genetic: Blood sample analysis — Nucleic acids sequencing, presence of proteins and metabolites.
Other: Health status — Health status will be examined by a physician and subject will complete a health status questionnaire.
Other: Race and ethnicity — Subject will complete race and ethnicity questionnaire to make sure subjects are from the Czech population.

SUMMARY:
This study will determine reference genomic, transcriptomic, proteomic and metabolomic profiles in Czech population and will evaluate its correlation with the disease phenotype.

DETAILED DESCRIPTION:
This study will determine reference genomic, transcriptomic, proteomic and metabolomic profiles in Czech population. Initially, there will be 1000 healthy volunteers, with the planned expansion to 10.000 participants (healthy volunteers and patients with different types of disease). Formation of the reference database of healthy volunteers and their parameters will allow a correct interpretation of the potential pathological findings in patients. It is very important to obtain healthy controls from the region of the Czech Republic, Central Europe respectively; since it is not possible to reliably compere ethnically and geographically diverse populations, which have generated in a different context and where the diseases manifest with other etiology ad phenotype. Although, in the limited measure, the similar molecular data exist in foreign databases, these are not compiled from the inhabitants of the Czech Republic, Central Europe not even from Slavic population. Study participants may volunteer for archiving of remaining biological materials for future studies.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 68 years
* (for the first 1100 subjects):
* healthy volunteers without genetically dependent disease and without such a disease in a family
* healthy volunteer without the preliminary evidence of civilizational diseases such as hypertension, diabetes, autoimmune and tumor diseases or acute infectional diseases; clinically manifesting cardiovascular or pulmonary disability.
* subject without permanent of long-term medication in the time of biological sampling.

Exclusion Criteria:

* not complying with inclusion criteria

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Selection from the blood donnors from the blood transfusion department.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Whole Genome (Exom) Sequencing of the Healthy Volunteers - establishment of the HEALTHY VOLUNTEER REFERENCE GENOME (min. 1000 individuals) | 72 months
  Establishment of the Healthy Volunteers Whole Genome (Exom) Reference Database typical for the population of the Czech Republic/Central Europe.
Whole Genome (Exom) Sequencing of the patient groups with different diseases and their comparison to the HEALTHY VOLUNTEER REFERENCE GENOME | 72 months
  Whole Genome (Exom) Sequencing of the patient populations presenting various diseases. Based on the comparison with the HEALTHY VOLUNTEER REFERENCE GENOME - determination of various genetic polymorphisms (single nucleotide polymorphisms, insertions, deletions, inversions, copy-number variations etc.) and giving these into correlation with disease phenotypes.

SECONDARY OUTCOMES:
Evaluation of the correlation with the disease phenotype | 72 months
  Based on the reference database of healthy volunteers in the Czech Republic a potential correlations will be evaluated among genomic, proteomic and metabolomic profiles of patients and the disease phenotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Marian Hajduch, MD, PhD., Study Director — IMTM, Palacky University in Olomouc, Faculty of Medicine and Dentistry
Locations (1):
- University Hospital Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: No